CLINICAL TRIAL: NCT02883075
Title: Measurement of Hemodynamic Variables Under Spinal Anesthesia in a Patient Undergoing Cesarean Section With Varied Positioning - a Comparative Study
Brief Title: Measurement of Hemodynamic Variables Under Spinal Anesthesia With Varied Positioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB #16-0119
Record Dates: First submitted 2016-07-21; First posted 2016-08-30 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2018-11

CONDITIONS: Pregnancy; Anesthesia
MeSH Terms: interventions — Supine Position

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supine position (Sham Comparator): Supine position Supine position after placement of spinal anesthetic
  Interventions: Other: Supine position
- Right lateral position (Active Comparator): Right lateral position Right lateral after placement of spinal anesthetic
  Interventions: Other: Right lateral position
- Left lateral position (Active Comparator): Left lateral position Left lateral after placement of spinal anesthetic
  Interventions: Other: Left lateral position

INTERVENTIONS:
Other: Supine position — Spinal anesthesia in sitting position then 2 minutes in Supine position after spinal anesthetic administration
  Arms: Supine position
Other: Right lateral position — Spinal anesthesia in sitting position then 2 minutes in the right lateral position after spinal anesthetic administration
  Arms: Right lateral position
Other: Left lateral position — Spinal anesthesia in sitting position then 2 minutes in the left lateral position after spinal anesthetic administration
  Arms: Left lateral position

SUMMARY:
Multiple studies have compared spinal anesthetic performed supine versus lateral, with varying results, in parturients having elective cesarean section. Needle positioning during spinal placement has also been examined. No positioning techniques have demonstrated definitive superiority for hemodynamic stability.

Investigators propose that following spinal placement in the sitting position if the patient is placed in a lateral position for 90 seconds prior to turning them supine, hemodynamic changes caused by sympathectomy related to the subarachnoid block can be avoided.

This is the first study to examining the influence of position changes after spinal anesthetic placement in the sitting position, which includes hemodynamic variables not previously studied including cardiac output, TPR (total peripheral resistance) and pulse pressure variation (PPV).

DETAILED DESCRIPTION:
Cesarean section is chosen when natural spontaneous vaginal delivery is either not possible or when the health of the baby or mother is compromised. Cesarean section may be planned, urgent, or performed emergently when the life of the baby or mother is threatened.

Cesarean section is performed using different anesthetic techniques including: spinal, epidural, combined spinal and epidural, and general anesthesia. Spinal anesthesia is the most common technique chosen due to its relative safety, rapid onset and avoidance of potential complications from general anesthesia. It is the technique of choice for elective cesarean section unless contraindicated. Spinal anesthesia causes sympathetic blockade followed by sensory and motor blockade. Nerve fiber size explains the speed of onset and differential block. The critical moments during spinal anesthesia come as soon as local anesthetic is injected into the subarachnoid space.

ELIGIBILITY:
Inclusion Criteria:

* Parturients undergoing elective cesarean section under spinal anesthesia
* Singleton intrauterine pregnancy with appropriate gestational age fetus (AGA) at gestational age 37 to 42 weeks

Exclusion Criteria:

* Large for gestational age, small for gestational age, and multiple gestations
* Patients with cardiovascular disease like hypertension, etc.
* Non-English or non-Spanish speakers
* BMI >40
* Inadequate or failed blocks and inadvertently high levels of spinal blockade will be dropped from the study
* Incarcerated parturients
* Expected heavy bleeding (placenta accreta, vascular anomaly, etc.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-11-26 (Actual)

PRIMARY OUTCOMES:
Heart rate | Immediately before spinal anesthestic placement through placental delivery
  Continuous Heart rate (beats per minute) measurements.
Blood pressure | Immediately before spinal anesthetic placement through placental delivery
  Continuous Blood pressure (mmHg) measurements

SECONDARY OUTCOMES:
Incidence of nausea and vomiting | Number of events spinal anesthetic placement through placental delivery
  Nausea and vomiting incidence and anti-emetic administration with time stamps will be documented.
Anti-emetic medication | Number of events spinal anesthetic placement through placental delivery
  Anti-emetic administration with time stamps will be documented.
Incidence of vasopressor usage | Spinal anesthetic placement through placental delivery
  Number of vasopressor use events will be monitored and recorded.
Total vasopressor usage | Spinal anesthetic placement through placental delivery
  All vasopressor administrations with time stamps will be documented.
Non Invasive Cardiovascular measurements: cardiac output | Spinal anesthetic placement through placental delivery
  Continuous Cardiac output (L/min) measurements
Non Invasive Cardiovascular measurements: stroke volume | Spinal anesthetic placement through placental delivery
  Continuous Stroke volume (mL) measurements
Non Invasive Cardiovascular measurements: TPR (total peripheral resistance) | Spinal anesthetic placement through placental delivery
  Continuous TPR (total peripheral resistance, dynes*sec/cm3)measurements

CONTACTS AND LOCATIONS:
Overall Officials: Ranganathan Govindaraj, MD, FRCA, Principal Investigator — The University of Texas Medical Branch, Galveston
Locations (1):
- UTMB, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No